CLINICAL TRIAL: NCT07309614
Title: A Multinational, Investigator-initiated, Parallel Group, Randomised, Double-blind, Placebo-controlled Phase 3b Superiority Trial Assessing the Effect of Dupilumab on Inducing Clinical Remission Outcomes in At-risk Type-2 Inflammatory Asthma (HOTHOT)
Brief Title: A Study Assessing the Effect of Dupilumab on Inducing Clinical Remission in Asthma
Acronym: HOTHOT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Sanofi (Industry); University of Oxford (Other); The University of Western Australia (Other); Regeneron Pharmaceuticals (Industry); Fonds de la Recherche en Santé du Québec (Other Government); Association Pulmonaire du Quebec (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024ESR0000238
Record Dates: First submitted 2025-11-25; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Asthma Control
Keywords: Asthma; Asthma control; moderate asthma; dupilumab; remission; type-2 inflammation; blood eosinophils; feno; exacerbations; trial; RCT
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Double blinded study assessing intervention versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Injection
- Dupilumab (Experimental)
  Interventions: Drug: Dupilumab Prefilled Syringe

INTERVENTIONS:
Drug: Dupilumab Prefilled Syringe — Dupilumab 400mg subcut x1 followed by 200mg subcut every 2 weeks
  Arms: Dupilumab
Drug: Placebo Injection — Volume-matched placebo injected subcut every 2 weeks
  Arms: Placebo

SUMMARY:
This study tests whether an asthma medication called dupilumab can help people achieve complete asthma control (called "remission") when given earlier in their disease, before asthma becomes severe. Currently, most people with asthma only receive advanced treatments like biologics after their condition has worsened significantly and caused lung damage. This study explores whether treating high-risk patients earlier could prevent asthma attacks and lung function decline, potentially achieving remission before permanent damage occurs. The study is looking for adults aged 18-79 with moderate asthma who have had at least one asthma attack requiring steroid pills in the past 2 years, use medium or high-dose inhaled steroids regularly, have high levels of inflammation markers in their blood and breath tests, but don't yet meet criteria for severe asthma requiring biologic therapy. Participants receive either dupilumab or placebo injections every 2 weeks for one year, alongside their regular asthma medications. They attend clinic visits every 3 months for breathing tests, questionnaires, and safety monitoring. Neither participants nor doctors know who receives the real medication until the study ends. The goal is to learn whether early treatment with dupilumab helps more people achieve complete asthma control compared to standard care alone, potentially changing how asthma is treated from "waiting until severe" to "preventing severe disease." The study runs in Canada, the United Kingdom, and Australia, involving 150 participants

DETAILED DESCRIPTION:
Asthma is a prevalent chronic respiratory disease for which 44% of people require oral corticosteroids (OCS) every year 1 . Whilst asthma is still managed on a damage-based schema allowing for unacceptable toxicities and irreversible airway remodelling, dupilumab and other type-2 targeting biologics have taught us that people with the highest type-2 inflammatory burden can achieve life-changing responses 2-6 . The term 'remission' has been used to describe the best possible outcome with biologics 5 . Across studies and molecules, remission was more likely to be achieved in people with shorter disease duration, lower morbidity, and higher type-2 inflammatory biomarkers 5,7-9 . These observations have increased interest in the earlier use of biologics in a Predict and Prevent framework 5,10-12 .

The HOTHOT study is a double-blind, placebo-controlled study assessing the effect of dupilumab on induction of clinical remission outcomes in type-2 high patients recruited before they develop severe uncontrolled asthma meeting current biological treatment recommendations. Dupilumab will be compared with placebo in 150 patients undergoing traditional symptom-based inhaled corticosteroid (ICS) up- and down-titration (as per current asthma guidelines). The target population is at-risk type-2 high asthma, defined as at-least medium-dose ICS, with a previous history of a systemic corticosteroid (SCS)-treated asthma attack in the last 24 months and blood eosinophils ≥ 0.3×109/L plus exhaled nitric oxide ≥35 ppb. These inclusion criteria are unique because they will target people with asthma who are at risk of severe asthma attacks and lung function decline, also not meeting current biological prescription/reimbursement criteria. The one-year active treatment adjustment period of the study will test the hypothesis that remission outcomes are more likely to be achieved with early targeted intervention with dupilumab compared to traditional symptom-guided management, where ICS up- and down-titration occurs independently of the presence of type-2 inflammation. The primary outcome, the win ratio based on remission criteria, assesses the likelihood of achieving remission 'wins' based on a hierarchy of criteria, while the secondary remission multi-component (yes/no) outcome, a binary (yes/no) multi-component endpoint for remission, offers a straightforward and comprehensive measure. The primary and secondary remission outcome measurements are both powered to be statistically and clinically impactful to move the need forward in the field of asthma. If correct, the hypothesis that earlier intervention with dupilumab significantly induces remission will shift the treatment paradigm from the usual 'wait and react' approach to a proactive risk-based 'predict and prevent' intervention using earlier targeted therapy in at-risk type-2 inflammatory disease.

ELIGIBILITY:
INCLUSION CRITERIA

Study participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Participant must be 18-<80 years of age at the time of signing the informed consent.

   Type of participant and disease characteristics
2. Physician diagnosis of asthma (according to GINA 2025) for ≥6 months, with documented historical airflow variability by one of the following:

   * Positive reversibility test: ≥12% and 200 ml in FEV1 after SABA administration at any point prior to randomisation
   * Airflow variability in clinic FEV1 >12% and 200 mL between historical clinical visits
   * Positive bronchial challenge test: fall in FEV1 of ≥20% with standard doses of methacholine (<16 mg/mL or <400mcg); or ≥10% with standardised hyperventilation, or exercise challenge test; or ≥15% with hypertonic saline or mannitol challenge
   * Peak flow variability of >20% between two assessments
3. Evidence of elevated type-2 biomarkers defined as both of:

   1. peripheral BEC ≥ 0.3×109/L at screening visit
   2. FeNO ≥ 35 ppb at screening visit
4. At least 1 asthma attack in the last 2 years, defined as acute asthma requiring SCS for ≥ 3 days or an emergency/hospital visit requiring SCS.
5. Treatment and evident adherence to a stable at-least medium-dose ICS (fluticasone propionate equivalent >250 mcg/day) for at least 3 months (including run-in period) [additional controllers e.g. LABA, LAMA or LTA are allowed]. The ICS dosage will be defined as the dosage received on a regularly basis, excluding extra reliever doses taken in the context of anti-inflammatory reliever (AIR) therapy from the calculation. AIR is allowed in the context of the study. Thus, the high-dose ICS trial population (fluticasone propionate equivalent >500 mcg/day)* will represent patients who are not meeting the exacerbation criteria for biological reimbursement.

   *As per section 6.2, we will cap recruitment to 60% of target population on medium-dose ICS, 40% on high-dose ICS, with randomisation also stratified by these categories.
6. Presence of one (or more) of the following additional risk factors for asthma attacks32 at screening or baseline: (i) uncontrolled asthma symptoms indicated by ACQ5 score of ≥ 1.5; (ii) impaired lung function indicated by post-bronchodilator FEV1 of ≤ 80% predicted; (iii) high-dose maintenance ICS therapy (iv) severe asthma attack in past 1-<12 months.

   Sex, contraceptive/barrier method and pregnancy testing requirements
7. Female participants

   a. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   i. Is a woman of nonchildbearing potential (WONCBP) as defined in the Study Manual.

   OR ii. Is a WOCBP and agrees to use a contraceptive method that is highly effective, with a failure rate of <1%, during the intervention period (to be effective before starting the intervention) and for at least 12 weeks after the last dose of study intervention.

   b. A WOCBP must have a negative highly sensitive serum pregnancy test at V1 (screening visit) and urine or serum pregnancy test (as required by local regulations) on Day 1 before the first dose of study intervention, c. If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

   d. Additional requirements for pregnancy testing during and after study intervention are imposed.

   e. The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a female participant with an early undetected pregnancy.

   Informed consent
8. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

4.2 EXCLUSION CRITERIA

Participants are excluded from the study if any of the following criteria apply:

Medical conditions

1. Use of SCS < 1 months prior to screening or on maintenance SCS.
2. Current tobacco smoker or recently stopped smoker (<6 months)
3. Ex-smoker with greater than 10 pack-years AND post bronchodilator FEV1/FVC ratio below the lower limit of normal according to GLI race-neutral standards. 69
4. Documented nonadherence to ICS, defined as dispensing of less than 75% of the prescribed ICS dose over the past 12 months (or annualised if less than 12 months), based on pharmacy refill records checked at screening.
5. Presence of significant and uncorrectable inhaler technique deficiencies, as assessed by the research team during inhaler technique evaluation at screening.
6. Contra-indication to study drug
7. Immunological disease, condition or medication that may affect the inflammatory response according to Investigator.
8. History of other significant lung disease e.g. lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, clinically significant bronchiectasis, chronic obstructive lung disease, or Churg-Strauss.
9. Severe concomitant illness (including known or suspected immunodeficiency) that, in the Investigator's judgement will adversely affect the participant's participation in the study.
10. Active malignancy or history of malignancy within 5 years (except for basal cell carcinoma of the skin).
11. Exposure to monoclonal antibody therapy for asthma or another investigational medicinal product within 5 half-lives of the drug.
12. Eligibility to Dupilumab based on licensed and reimbursed indications in the participant's jurisdiction (e.g. nasal polyposis, atopic dermatitis, eosinophilic esophagitis, prurigo nodularis, etc.)
13. Treatment with live (attenuated) vaccine in the past 4 weeks.
14. Prohibited medication

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Win ratio based on remission criteria | Week 4 to Week 56 (except FEV1 change: Week 0 values serve as baseline)
  Win ratio comparing patients achieving clinical remission outcomes in dupilumab group vs placebo group, based on remission criteria.
  The unmatched paired testing will follow this hierarchy:
  1. Study participant has not had a severe asthma attack between weeks 4 and 56
  2. Number of asthma attacks between weeks 4 and 56
  3. Improved or stable lung function (defined as a decline from parent study baseline in pre- or postbronchodilator FEV1 by no more than 5%) at Week 56
  4. No more than medium-dose ICS maintenance therapy (as defined by GINA 2025) at Week 56
  5. 5-item Asthma Control Questionnaire mean score <1.5 at Week 56

SECONDARY OUTCOMES:
Annualised severe asthma attack rate | Week 4 to Week 56
  Reduction in annualised severe asthma attack rate with dupilumab vs placebo
Win ratio for clinical remission in medium-dose ICS subgroup | Week 4 to Week 56 (except FEV1 change: Week 0 values serve as baseline)
  Win ratio comparing remission outcomes in dupilumab vs placebo among patients on medium-dose ICS at enrolment.
  The unmatched paired testing will follow this hierarchy:
  1. Study participant has not had a severe asthma attack between weeks 4 and 56
  2. Number of asthma attacks between weeks 4 and 56
  3. Improved or stable lung function (defined as a decline from parent study baseline in pre- or postbronchodilator FEV1 by no more than 5%) at Week 56
  4. No more than medium-dose ICS maintenance therapy (as defined by GINA 2025) at Week 56
  5. 5-item Asthma Control Questionnaire mean score <1.5 at Week 56
Change in FEV1 postbronchodilator | Week 0 to Week 56
  Change in FEV1 postbronchodilator (L) with dupilumab vs placebo
Proportion of patients achieving clinical remission at 1 year | Week 4 to Week 56 (except FEV1 change: Week 0 values serve as baseline)
  Proportion of patients achieving clinical remission at 1 year in dupilumab vs placebo group
  Study participants meet ALL of the follow criteria at Week 56:
  1. Study participant has not had a severe asthma attack between weeks 4 and 56
  2. Improved or stable lung function (defined as a decline from parent study baseline in pre- or postbronchodilator FEV1 by no more than 5%) at Week 56
  3. No more than medium-dose ICS maintenance therapy (as defined by GINA 2025) at Week 56
  4. ACQ5 <1.5 at Week 56
Effect of dupilumab on corticosteroid use, compared to placebo | Week 0 to Week 56
  Cumulative prescribed dose of systemic corticosteroids (prednisone-equivalent mg)
Effect of dupilumab on asthma symptoms, compared to placebo | Week 0 to Week 56
  Change from in 5-item Asthma Control Questionnaire (mean score). The score ranges from 0 to 6 : higher scores indicate worse asthma control.
Effect of dupilumab on absenteism, compared to placebo | Week 0 to Week 56
  Cumulative time off work or education due to asthma symptoms
Effect of dupilumab on unplanned healthcare attendencances, compared to placebo | Week 0 to Week 56
  Cumulative number of unplanned healthcare attendances
Effect of dupilumab on emergency room attendance, compared to placebo | Week 0 to Week 56
  Cumulative number of emergency department visits
Effect of dupilumab on hospilisation use, compared to placebo | Week 0 to Week 56
  Cumulative number of hospitalisations
Effect of dupilumab on asthma-related quality of life, compared to placebo | Week 0 to Week 56
  Change in Asthma Quality of Life Questionnaire with Standardised Activities AQLQ(S). The score ranges from 1 to 7 : higher scores indicate better quality of life.
Effect of dupilumab on respiratory disease-related quality of life, compared to placebo | Week 0 to Week 56
  Change in Saint-George Respiratory Questionnaire. The score ranges from 0 to 100 : higher scores indicate worse health status.
Effect of dupilumab on health-related quality of life, compared to placebo | Week 0 to Week 56
  Change in health-related quality of life questionnaire EQ-5D. The index value typically ranges from approximately -0.59 to 1.0: higher values indicate better health related quality of life.
Effect of dupilumab on work and activity productivity, compared to placebo | Week 0 to Week 56
  Change in Work Productivity and Activity Impairment Score for asthma (WPAI-Asthma). The score ranges from 0 to 100 percent: higher values indicate greater impairment or worse outcomes.
Effect of dupilumab on maintenance ICS dose, compared to placebo | Week 0 to Week 56
  Change in maintenance ICS dose (continuous and categorical: very low, low, medium, high-dose , as per GINA 2025)
Effect of dupilumab on type-2 biomarkers, compared to placebo | Week 0 to Week 56
  Change in blood eosinophil count, FeNO, and IgE levels, expressed as % relative to baseline
Effect of dupilumab on reported usage of reliever medication, compared to placebo | Week 0 to Week 56
  Change in reported usage of reliever medication (mean reliever use per week)
Effect of dupilumab vs placebo on sino-nasal symptoms | Week 0 to Week 56
  Change in Sino Nasal Outcome Test 22 score. The score ranges from 0 to 110 : higher scores indicate worse symptom severity.

OTHER OUTCOMES:
To describe exacerbation phenotypes and SCS-responsiveness in the dupilumab and placebo arms. | Pre- (day 1 of exacerbation, pre-treatment) and Post-treatment visit (day 7)
  Change in FEV1 post-BD (L) following SCS treatment
To evaluate safety of dupilumab in this population of patients | Week 0 to Week 56
  Incidence of treatment-emergent adverse events (TEAE) and serious adverse events (SAE) in treatment group vs placebo

CONTACTS AND LOCATIONS:
Locations (5):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- Canada (3):
  - McGill University Health Centre, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - CIUSSS de l'Estrie- CHUS, Sherbrooke, Quebec
- Oxford University Hospitals NHS Foundation Trust - John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the time of publication of the study results, the REDCap data dictionary, analytical code used to process the data, and analytical code used to analyze the outcomes will be posted on Github.
  In addition, after the end of the study, the data collected as part of the study can be shared as follows:
  • A copy of the coded data collected as part of the study and under the control of the sponsor will be created and all data will be :
  * Anonymized and the sponsor will ensure to the fullest extent possible that the data irremediably no longer allows any study participant to be identified directly or indirectly; or
  * Subject to additional de-identification process to remove additional identifiers to ensure that the data no longer allows the study participants to be directly identified; Following that process, the anonymized/further deidentified dataset could be shared with the participating sites and their respective investigators for their own internal and non-commercial uses in accordanc
Supporting Information: Study Protocol, SAP, CSR, Analytic Code